CLINICAL TRIAL: NCT04429542
Title: First-in-Human, Phase 1/1b, Open-label, Multicenter Study of Bifunctional EGFR/TGFβ Fusion Protein BCA101 Monotherapy and in Combination Therapy in Patients With EGFR-Driven Advanced Solid Tumors
Brief Title: Study of Safety and Tolerability of BCA101 Monotherapy and in Combination Therapy in Patients With EGFR-driven Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Bicara Therapeutics (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BCA101X1101; KEYNOTE-E28 (Other: Merck Sharp & Dohme LLC)
Record Dates: First submitted 2020-06-10; First posted 2020-06-12 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Head and Neck Squamous Cell Carcinoma; Squamous Cell Carcinoma of Anal Canal; Colorectal Cancer; Squamous Cell Carcinoma of the Lung; EGFR Amplification; Epithelial Ovarian Cancer; Pancreas Cancer; Cutaneous Squamous Cell Carcinoma; Head and Neck Neoplasms; Carcinoma, Squamous Cell; Squamous Cell Carcinoma of Head and Neck
Keywords: TGFβ; EGFR; pembrolizumab; ficerafusp alfa
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Colorectal Neoplasms; Carcinoma, Ovarian Epithelial; Pancreatic Neoplasms; Head and Neck Neoplasms; Carcinoma, Squamous Cell | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- BCA101 Monotherapy (Experimental): Route: IV Infusion Frequency: QW Current Dose: 1500mg
  Interventions: Drug: BCA101
- BCA101 + pembrolizumab (Experimental): Route: IV Infusion Frequency: Q3W Dose: 200mg
  Interventions: Drug: BCA101; Drug: Pembrolizumab

INTERVENTIONS:
Drug: BCA101 — EGFR/TGFβ fusion monoclonal antibody
  Other Names: Ficerafusp alfa
Drug: Pembrolizumab — anti-PD-1
  Arms: BCA101 + pembrolizumab

SUMMARY:
The investigational drug to be studied in this protocol, BCA101, is a first-in-class compound that targets both EGFR with TGFβ. Based on preclinical data, this bifunctional antibody may exert synergistic activity in patients with EGFR-driven tumors.

DETAILED DESCRIPTION:
This is a Phase 1/1b, open-label study, which consists of dose escalation parts (Part A) followed by expansion cohorts (Part B) for both single agent BCA101 and combination BCA101 plus pembrolizumab.

The study population in dose escalation (Part A) of single agent BCA101 consists of subjects with EGFR-driven advanced solid tumors refractory to standard of care or for whom no standard of care is available. Dose escalation (Part A) of combination BCA101 and pembrolizumab consists of subjects with either Squamous Cell Carcinoma of the Head and Neck (HNSCC) or Squamous Cell Carcinoma of the Anal Canal (SCCAC) whose tumors are refractory to standard of care or for whom no standard of care is available.

Once the maximum tolerated dose (MTD) / recommended dose (RD) of single agent BCA101 is determined, the study will continue with expansion cohorts (Part B) with select tumor types. Expansion cohorts for single agent BCA101 will include cutaneous squamous cell carcinoma. Planned expansion cohorts for the combination of BCA101 and pembrolizumab include: 1) HNSCC and 2) SCCAC.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have measurable disease amendable to biopsy and be willing to undergo both a pre-treatment and on-treatment biopsy, as well as provide archival tumor if available from the primary tumor (a paraffin embedded tumor tissue block sufficient to obtain at least 10 sections of 4 to 5 micrometer thickness).
* Patient must have a performance status of ≤1 on the Eastern Cooperative Oncology Group Performance Scale.
* Patients must have evaluable or measurable disease (computed tomography [CT]/magnetic resonance imaging [MRI] scans performed within 21 days before the screening visit are acceptable) demonstrating measurable disease, i.e., at least 1 unidimensional measurable lesion as defined by Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST 1.1) and Immune Response Evaluation Criteria in Solid Tumors (iRECIST).
* Tumor eligibility:

PART B (Cohort expansion):

1. Single agent BCA101 - patients with the following tumor type will be eligible:

   • Expansion Cohort 1: Cutaneous Squamous Cell Carcinoma (CSCC) - i. patients must have received (or been intolerant to or ineligible for) prior anti-PD-1 therapy in the metastatic or locally advanced setting.

   ii. No prior history of treatment with anti-EGFR antibodies in the unresectable/metastatic setting (prior treatment with radiotherapy in the adjuvant setting is allowed).
2. Combination BCA101 and pembrolizumab - patients with the following tumor types will be eligible:

   • Expansion Cohort 2: Head and Neck Squamous Cell Carcinoma (HNSCC), metastatic or unresectable, recurrent with a Combined Positive Score (CPS) equal to or greater than 1, as determined by an CLIA-approved laboratory test. Primary tumor locations of oropharynx, oral cavity, hypopharynx, or larynx. Participants may not have a primary tumor site of nasopharynx (any histology).

   i. Patients must have no prior systemic therapy administered in the recurrent or metastatic setting (with the exception of systemic therapy completed >6 months prior if given as part of multimodal treatment for locally advanced disease) or prior history of immune checkpoint inhibitors with the exception of neoadjuvant therapy (>6 months prior to study drug initiation). No prior history of anti-EGFR antibodies (with the exception of radiosensitizing agents and multimodal treatment for locally advanced disease).

   ii. Patients must provide tissue for PD-L1 biomarker analysis from a core or excisional biopsy (fine needle aspirate is not sufficient): A newly obtained biopsy (within 90 days prior to start of study treatment) is preferred but an archival sample is acceptable.

   iii. Patients must have results from testing of human papillomavirus (HPV) status for oropharyngeal cancer
   * Expansion Cohort 3: Squamous Carcinoma of the Anal Canal (SCAC), locally advanced/unresectable or metastatic.

     i. Patients must have received (or been intolerant to or ineligible for) at least 1 prior line of chemotherapy and received no more than 2 prior lines of systemic treatments for treatment of unresectable and/or metastatic disease. No prior history of immune checkpoint inhibitors.
   * Expansion Cohort 5: Squamous Non-Small Cell Lung Cancer (SqNSCLC) i. Patients must have a histologically or cytologically confirmed diagnosis of stage IV (AJCC 8th edition) squamous NSCLC. Patients with mixed histology (e.g., adenosquamous) are not allowed.

   ii. Patients must have progressed on one prior systemic therapy in the metastatic setting.

   iii. No prior history of treatment with anti-EGFR antibodies in the metastatic setting.

   • Expansion Cohort 6: Head and Neck Squamous Cell Carcinoma (HNSCC), metastatic or unresectable, recurrent with a Combined Positive Score (CPS) less than 1, as determined by PD-L1 IHC 22C3 pharmDx.
3. Randomized to either ficerafusp alfa alone or in combination with pembrolizumab • Expansion Cohort 9: Colorectal cancer (CRC) i. Patients must have received at least 2 and no more than 3 prior lines of systemic therapy including two standard treatment regimens.

Exclusion Criteria:

* For Part A: Exposure to anti-EGFR antibodies within 4 weeks of the first dose of study drug.
* Prior treatment with any anti-TGFβ therapy.
* Prior history of Grade ≥ 2 intolerance or hypersensitivity reaction to cetuximab or other anti-EGFR therapy or other murine proteins or prior discontinuation of therapy in the setting of toxicity related to treatment.
* Pregnant or breastfeeding women.
* Any condition requiring systemic treatment with either corticosteroids (>10 mg daily of prednisone or equivalent) or other immunosuppressive medication within 14 days prior to the first dose of study drug, with the exception of topical, intranasal, intrabronchial, or ocular steroids.
* Known history of a hematologic malignancy (or solid tumor other than the ones indicated for this study), unless the patient has undergone potentially curative therapy with no evidence of that disease for 2 years. Does not include tumors with a negligible risk of metastasis or death (e.g. adequately treated basal or squamous cell carcinoma, stage 1 prostate cancer, or carcinoma in situ of the cervix or carcinoma in situ of the breast). Subjects enrolling in the CSCC cohort may have chronic lymphocytic leukemia as long as the patient is not on active treatment.
* Known cases of human immunodeficiency virus (HIV) are excluded if patients have a CD4+ T-cell (CD4+) count <250 cells/uL. To ensure that effective antiretroviral therapy (ART) is tolerated and that toxicities are not confused with investigational drug toxicities, trial participants should be on established ART for at least four weeks and have an HIV viral load less than 400 copies/mL prior to enrollment.
* Patients with chronic HBV infection with active disease who meet the criteria for anti-HBV therapy and are not on a suppressive antiviral therapy prior to initiation of study treatment
* Patients with a known history of hepatitis C who have not completed curative antiviral treatment or have a HCV viral load above the limit of quantification

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 292 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Safety of BCA101 alone and BCA101 in combination with pembrolizumab: Incidence and severity of AEs and SAEs | 24 months
  Incidence and severity of AEs and SAEs
Tolerability of BCA101 alone and BCA101 in combination with pembrolizumab: Incidence and severity of AEs and SAEs | 24 months
  Incidence and severity of AEs and SAEs
Incidence of Dose Limiting Toxicities (DLTs) | 21 days
  Incidence of DLTs during the first cycle of treatment with BCA101 monotherapy or the combination of BCA101 and pembrolizumab.

SECONDARY OUTCOMES:
Objective Response Rate | 24 months
  Determine objective response rate in each part of the study, per RECIST v1.1 and iRECIST
Clinical Benefit Rate | 24 months
  Determine clinical benefit rate in each part of the study, per RECIST v1.1 and iRECIST
Progression free survival | 24 months
  Determine PFS in each part of the study, per RECIST v1.1 and iRECIST
Duration of Response | 24 months
  Determine duration of response in each part of the study, per RECIST v1.1 and iRECIST
Overall Survival | 24 months
  Determine survival rates in each part of the study.
AUC of BCA101 and pembrolizumab | 24 months
  AUC
Cmax of BCA101 and pembrolizumab | 24 months
  Cmax
Tmax of BCA101 and pembrolizumab | 24 months
  Tmax
Concentration vs time profile of BCA101 and pembrolizumab | 24 months
  Ctrough
Half-life of BCA101 and pembrolizumab | 24 months
  Half-life
Immunogenicity of BCA101 and pembrolizumab | 24 months
  Incidence and titer of anti-drug-antibodies

CONTACTS AND LOCATIONS:
Locations (20):
- United States (15):
  - Moores Cancer Center UC San Diego Health, La Jolla, California
  - Keck School of Medicine of USC, Los Angeles, California
  - UCLA, Los Angeles, California
  - University of California, Davis Comprehensive Cancer Center, Sacramento, California
  - H. Lee Moffitt Cancer Center and Research Institute, Inc, Tampa, Florida
  - Dana Farber/Partners Cancer Care Inc, Boston, Massachusetts
  - Memorial Sloan Kettering, New York, New York
  - Columbia University Herbert Irving Comprehensive Cancer Center, New York, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Hollings Cancer Center, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
- Australia (4):
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - Calvary Mater Newcastle, Waratah, New South Wales
  - Austin Hospital, Heidelberg, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No